CLINICAL TRIAL: NCT03369990
Title: A Randomized, Double-blind, Placebo-controlled, Phase Ⅱ Optimal Dose-finding Study to Determine the Safety and Efficacy of DWP450 in Subjects With Benign Masseteric Hypertrophy
Brief Title: DWP450 Treatment in Subjects With Benign Masseteric Hypertrophy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP450008
Record Dates: First submitted 2017-11-26; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Benign Masseteric Hypertrophy
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin type A (Experimental): DWP450
  Interventions: Drug: Botulinum toxin type A
- Placebo (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin type A(DWP450)
  Arms: Botulinum toxin type A
Drug: Placebos — Normal Saline
  Arms: Placebo

SUMMARY:
This study is A Randomized, Double-blind, Placebo-controlled, Phase II Optimal Dose-finding Study to Determine the Safety and Efficacy of DWP450 in Subjects with Benign Masseteric Hypertrophy

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject over 18 years of age and written informed consent is obtained.
2. Subject with Benign Masseter Hypertrophy
3. Subject who has Bisymmetry of masseter at visual assessment.
4. Subjects who meets thickness of Masseter muscle by ultrasonography.
5. Subjects who can and will comply with the requirements of the protocol.

Exclusion Criteria:

1. Diagnosis of Myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function
2. Subject who got any treatment, including double jaw surgery, laser, thread treatment etc. in 12 months.
3. Subject who had previously received botulinum toxin within 3 months prior to the study entry
4. Subject with known hypersensitivity to botulinum toxin
5. Subject who are pregnant or lactating or found pregnancy though the urine or sebum test or disagreed to avoid pregnancy during study period.
6. Subjects who are not eligible for this study at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Reduction amount of masseter muscle thickness | At 12 weeks
  Reduction amount of masseter muscle thickness by Ultrasonography

SECONDARY OUTCOMES:
Reduction amount of masseter muscle thickness | At 4,8,16 weeks
  Reduction amount of masseter muscle thickness by Ultrasonography
Reduction amount of lower face volume | At 4, 8, 12, 16 weeks
  Reduction amount of lower face volume by 3D digital imaging
Overall satisfaction of subject | At 4, 8, 12, 16 weeks
  Overall satisfaction of subject by questionnaire